CLINICAL TRIAL: NCT05563168
Title: Multicenter, Double-blind, Randomized, Placebo-controlled Study Evaluating Diltiazem in Combination With Standard Treatment in the Management of Patients Hospitalized With COVID-19 Pneumonia - A Phase IIB, Proof of Concept Study
Brief Title: Study Evaluating Diltiazem in Combination With Standard Treatment in the Management of Patients Hospitalized With COVID-19 Pneumonia
Acronym: DICOV
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the epidemiological situation has changed considerably.
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Signia Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL21_0855; 2021-004160-94 (EudraCT Number)
Record Dates: First submitted 2022-09-30; First posted 2022-10-03 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: Pneumonia, Viral; Diltiazem
MeSH Terms: conditions — COVID-19; Pneumonia, Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Of Care (SOC) + diltiazem (Experimental): Patients will receive the standard of care at the time of their inclusion in the trial and will also receive diltiazem (60mg 3 times a day) for 7 days.
  Interventions: Drug: DILTIAZEM TEVA 60 mg or placebo
- SOC + placebo (Placebo Comparator): Patients will receive the standard of care at the time of their inclusion in the trial and will also receive a diltiazem placebo (3 times a day) for 7 days
  Interventions: Drug: DILTIAZEM TEVA 60 mg or placebo

INTERVENTIONS:
Drug: DILTIAZEM TEVA 60 mg or placebo — DILTIAZEM TEVA 60 mg 3 times a day during 7 days + standard of care Or placebo 3 times a day during 7 days + standard of care.

SUMMARY:
SARS-CoV-2 infection is responsible for hypoxemic pneumonia, which is sometimes serious and associated with excess mortality. To date, with the exception of dexamethasone, which has shown clinical efficacy by reducing the mortality of infected patients, no other therapeutic strategy has demonstrated a curative clinical benefit, particularly in the initial stages facilitating viral eviction. .

Based on the mechanism of action and the available data, diltiazem, administered in the first days post-infection, could facilitate viral eradication in these patients through the stimulation of the innate immune response of cells of the infected respiratory epithelium, actor in the fight against SARS-CoV-2.

In this context, the investigators propose the DICOV trial, to demonstrate the ability of diltiazem to reduce the viral load more rapidly, in patients hospitalized for COVID-19 hypoxemic pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or over
* SARS-CoV-2 infection proven by RT-PCR on a nasopharyngeal sample within 72 hours prior to inclusion in the study
* Onset of symptoms of viral infection ≤ 7 days
* Hospitalization required due to hypoxemia (air saturation < 94% at rest)
* Presence of radiological pneumopathy (chest X-ray or non-enhanced thoracic CT)
* Patient affiliated to a social security scheme.
* Patient capable of giving free, informed and written consent.
* Patient with a history of SARS-CoV-2 infection may participate in the study, but this infection must not have occurred within the 3 months prior to his current hospitalization.
* Patient who has been vaccinated against SARS-CoV-2 can participate in the study (regardless of the number of doses)
* Patient not eligible for specific anti-COVID treatment authorized in France (MA or early access) and not part of the standard of care at the time of the study
* Female patient of childbearing age using effective contraception during study participation, the same applies to partners of childbearing age of male patients. Male patients must use condoms.

Exclusion Criteria:

* Need for hospitalization in intensive care unit at inclusion
* Patient with cognitive impairment, at the discretion of the investigator
* Pregnant woman (positive urine pregnancy test on inclusion) or breastfeeding
* Participation in another interventional study or being in the exclusion period from a previous study
* Patient on diltiazem therapy
* Contraindication to diltiazem

  * Hypersensitivity to diltiazem or to any of the excipients
  * Unaided sinus dysfunction
  * Unaided 2nd and 3rd degree atrioventricular blocks
  * Left ventricular failure with pulmonary stasis (cardiogenic edema)
  * Severe bradycardia (≤ 40 beats per minute)
  * In combination with: dantrolene infusion, pimozide, dihydroergotamine, ergotamine, nifedipine, ivabradine, beta blockers, antiarrhythmics, esmolol, fingolimod.
* Patient with renal, hepatic or cardiac insufficiency (at the discretion of the investigator)
* Hypersensitivity to mannitol
* Use of anti-COVID medications other than those offered in routine testing and care.
* Presence of hemodynamic instability, systolic blood pressure < 100 mmHg, presence of multi-visceral failure
* Prior respiratory pathology requiring oxygen therapy at the long-term and/or non-invasive ventilation
* Immunocompromised patients (organ transplant, allograft, under chemotherapy, under Rituximab or a history of Rituximab), for any other situation seek the advice of the coordinating investigator
* Patient under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 viral load decrease between D1 and D7 | At day 1 and day 7 post treatment initiation.
  Dosage of the standardized SARS-CoV-2 viral load on nasopharyngeal samples on day 1 and day 7 after treatment initiation.

SECONDARY OUTCOMES:
Time to clinical improvement | Within 28 days post-randomization
  Time to clinical improvement (in days), defined as the time from randomization to an improvement of at least 2 points on a 7-point ordinal scale
Overall survival | at day 28
  Percentage of patients who died between D1 and D28 of the start of treatment
SARS-CoV-2 viral load kinetics | Day 1, day 7, day 15, day 21 and day 28
  Kinetics of viral load decrease by dosage of the normalized SARS-CoV-2 viral load on nasopharyngeal samples
proportion of patients who are potential transfer candidates in intensive care | At Day 15
  Percentage of patients candidates for transfer to intensive care at Day 15 of the start of treatment
Tolerance of the study treatment | Within 28 days after treatment initiation
  Occurrence of adverse events, severe adverse events and premature discontinuation of study treatment
Duration of oxygen therapy | Within 28 days after treatment initiation
  Number of days the patient was put on oxygen therapy
Proportion of patients requiring assisted or non-invasive ventilation | Within 28 days after treatment initiation
  Percentage of patients requiring assisted or non-invasive ventilation
Duration of assisted or non-invasive ventilation | Within 28 days after treatment initiation
  Number of days the patient was put on assisted or non-invasive ventilation
Duration of hospitalization in intensive care unit | At day 28.
  Number of days spent in intensive care
Duration of hospitalization in intensive care unit | At day 90
  Number of days spent in intensive care. For patients still in intensive care on D28 this information will be collected on D90
Hospital length of stay | At day 28.
  Number of days spent in hospital
Hospital length of stay | At day 90
  Number of days spent in hospital. For patients still in intensive care on D28 this information will be collected on D90
Flow rate of oxygen used | Within 28 days after treatment initiation
  Maximum oxygen rate used
Extension of viral pneumonitis | Day 1, day 28
  Difference in extension of viral pneumonitis on comparative analysis scans performed at D1 and D28

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Devouassoux, Pr, Principal Investigator — Departement of Pulmonology, Croix-Rousse Hospital, Hospices Civils de Lyon
Locations (21):
- France (21):
  - respiratory department Amiens Hospital, Amiens
  - Service de Maladies infectieuses et tropicales, Amiens
  - Département de Pneumologie, CHU Angers, Angers
  - Service de Pneumologie, CHU Besançon, Besançon
  - Service de pneumologie Hôpital Haut-Leveque, Bordeaux
  - Service de Pneumologie CHU Gabriel Montpied, Clermont-Ferrand
  - Service des Maladies Infectieuses et Tropicales, Fort-de-France
  - Maladies infectieuses et Tropicales CHU Grenoble Rhône-Alpes, Grenoble
  - Departement of Pulmonology, Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon
  - Médecine Interne, Hôpital de la Croix- Rousse, HOSPICES CIVILS DE LYON, Lyon
  - Clinique des bronches, de l'allergie et du sommeil Hôpital Nord, Marseille
  - de Pneumologie Groupe Hospitalier du Havre Hôpital, Montivilliers
  - Pulmonology department CHU Montpellier, Montpellier
  - Service Pneumologie, Hôpital BICHAT, Paris
  - Service de Pneumologie, GHU APHP-Sorbonne Université, site Pitié Salpêtrière, Paris
  - Service de pneumologie, CHLS, Hospices Civils de Lyon, Pierre-Bénite
  - Médecine interne, CHMS, Hospices Civils de Lyon, Pierre-Bénite
  - Department of Pulmonology-Thoracic Oncology, University Hospital of SaintEtienne, Saint-Etienne
  - Service de pneumologie, CHRU Strasbourg, Strasbourg
  - Clinique des Voies Respiratoires Hôpital Larrey, Toulouse
  - Service des Maladies Infectieuses et du Voyageur Hôpital Gustave Dron, Tourcoing